CLINICAL TRIAL: NCT06561880
Title: A Multi-center, Single-arm Trial of the Efficacy of a Triple Regimen Including Gilteritinib, Venetoclax, and Azacitidine in Newly Diagnosed Fit AML Patients With FLT3 Mutation
Brief Title: The Efficacy of Triple Regimen in Newly Diagnosed AML Patients With FLT3 Mutation
Acronym: FLT3AML-2024
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024055
Record Dates: First submitted 2024-08-08; First posted 2024-08-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: FLT3 Gene Mutation; AML
MeSH Terms: interventions — gilteritinib; venetoclax; Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Triple Regimen Induction Including Gilteritinib, Venetoclax and Azacitidine (Experimental): Patients will receive 2 courses of induction with a triple regimen therapy consisting of Gilteritinib, Venetoclax, and Azacitidine. Patients who achieved complete remission will receive 3 courses of intermediate-dose cytarabine for consolidation. After consolidation therapy, dose-adjusted triple regimen therapy including Gilteritinib, Venetoclax, and Azacitidine will be applied for 6 courses as maintenance treatment.
  Interventions: Drug: Gilteritinib; Drug: Cytarabine

INTERVENTIONS:
Drug: Gilteritinib — Induction therapy regimen(2 courses):
  triple regimen therapy: Azacitidine 75mg/m2/d d1-7; Venetoclax 100mg d1,200mg d2,400mg d3-28; Gilteritinib (as required at admission: 80 or 120mg) d1-28.
  dose-adjusted triple regimen therapy: Azacitidine 75mg/m2/d d1-5; Venetoclax 400mg d1-7; Gilteritinib (as required at admission: 80 or 120mg) d1-28.
  Patients with no remission after the first induction course will receive another course with triple regimen therapy; Patients with complete remission after the first induction course will receive another course of dose-adjusted triple regimen therapy.
  Other Names: Venetoclax; Azacitidine
Drug: Cytarabine — Consolidation therapy (3 courses):
  intermediate-dose cytarabine regimen :2g/m2 q12h d1-3, age < 60 years;1g/m2 q12h d1-3, age ≥60 years.
  If NGS detected FLT3 mutation before consolidation chemotherapy, gilteritinib will be added during the consolidation course at d4-17.
  Other Names: Gilteritinib
Drug: Gilteritinib — Maintenance treatment (6 courses):
  dose-adjusted triple regimen therapy:Azacitidine 75mg/m2/d d1-5; Venetoclax 400mg d1-7; Gilteritinib (as required at admission: 80 or 120mg) d1-28.
  Other Names: Venetoclax; Azacitidine

SUMMARY:
The FMS tyrosine kinase 3 (FLT3) gene mutation occurs in 30% of newly diagnosed AML patients, leading to a higher relapse rate and mortality rate. In the past, multi-drug combination chemotherapy regimens had limited efficacy in newly diagnosed AML patients with FLT3 mutations, especially in those with FLT3-ITD. However, the FLT3 inhibitors greatly improved the survival of AML patients with FLT3 mutations. Although several studies have focused on the effectiveness of FLT3 inhibitor combination therapy for FLT3-mutated AML, further studies are needed to determine the optimal regimen and dosage. A triple regimen consisting of Gilteritinib, Venetoclax, and Azacitidine had shown good efficacy in unfit newly diagnosed FLT3-mutated AML patients. This clinical trial aims to determine the optimal dosage of the triple regimen and investigate its efficacy in newly diagnosed fit FLT3-mutated AML patients. Besides, this trial will provide evidence for treatment decisions based on measurable residual disease in patients with the triple regimen.

DETAILED DESCRIPTION:
This stuay intends to conduct a multi-center, single-arm clinical study to explore the efficacy of the triple induction regimen consisting of Gilteritinib, Venetoclax, and Azacitidine in newly diagnosed FLT3 mutated AML patients who are suitable for intensive chemotherapy. The maximum dose of Gilteritinib that can be safely combined with Azacitidine and Venetoclax will be determined. Patients will receive 2 courses of a triple regimen therapy for induction and those who achieved complete remission will receive 3 courses of intermediate-dose cytarabine for consolidation. After consolidation therapy, dose-adjusted triple regimen therapy will be applied for 6 courses as maintenance treatment. Bone marrow morphology and minimal residual disease detected by flow cytometry and next-generation sequencing will be monitored during the treatment to provide evidence for treatment decisions. Response and survival of patients will be recorded to evaluate the efficacy of the triple regimen.

ELIGIBILITY:
Inclusion Criteria:

1. MDS/AML patients WHO meet AML and ICC definitions according to WHO (2022) or ICC standards (10%-20% of bone marrow naive cells) and have FLT3-TKD or ITD mutations detected by PCR or second-generation sequencing.
2. Age ≥15 years old, male or female.
3. The physical status assessment (ECOG-PS) of the Eastern Oncology Collaboration group was 0-2 points.
4. Pass the requirements of the following laboratory tests (performed within 7 days before treatment) :

1) Total bilirubin ≤ 1.5 times the upper limit of normal value (same age); 2) AST and ALT≤ 2.5 times the upper limit of normal value (same age); 3) Blood creatinine < 2 times the upper limit of normal (same age); 4) Myocardial enzymes < 2 times the upper limit of normal (same age); 5) Echocardiography (ECHO) was performed to determine the ejection fraction of the heart within the normal range.

Exclusion Criteria:

1. Acute promyelocytic leukemia with PML-RARA fusion gene
2. Acute myeloid leukemia with RUNX1-RUNX1T1 or CBFB-MYH11 fusion gene
3. Acute myeloid leukemia with BCR-ABL fusion gene
4. Have treated patients (those who have previously received induction chemotherapy but can receive hydroxyurea down-cell therapy).
5. Concurrent malignant tumors of other organs (those requiring treatment).
6. Active heart disease, defined as one or more of the following:

1) A history of uncontrolled or symptomatic angina; 2) Myocardial infarction less than 6 months after enrollment; 3) Have a history of arrhythmia requiring drug treatment or severe clinical symptoms; 4) Uncontrolled or symptomatic congestive heart failure (> NYHA level 2); 5) The ejection fraction is lower than the lower limit of the normal range. 7. Serious infectious diseases (uncured tuberculosis, pulmonary aspergillosis). 8. Those who were not considered suitable for inclusion by the researchers.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of gilteritinib | up to 3 months after enrollment of the first participants
  The maximum dose of gilteritinib that can be safely combined with azacitidine and venetoclax
Event-free survival (EFS) | up to 2 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of failed to achieve complete remission, the date of relapse, or the date of death, whichever occurred first.
Complete remission (CR)/CR with partial hematologic recovery (CRh)/CR with incomplete hematologic recovery (CRi) with negative MRD detected by flow cytometry. | up to 1 years after the date of the last enrolled participants
  The ratio of CR/CRh/CRi with negative MRD detected by flow cytometry after induction, consolidation, and maintenance therapy.
CR/CRh/CRi with negative MRD detected by NGS (next-generation sequencing) | up to 1 years after the date of the last enrolled participants
  The ratio of CR/CRh/CRi with negative MRD detected by NGS after induction,consolidation, and maintenance therapy.

SECONDARY OUTCOMES:
CR/CRh/CRi rate | up to 3 months after the date of the last enrolled participants
  The ratio of patients achieved CR/CRh/CRi after two course of induction therapy
overall survival | up to 2 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of death or the date of last follow-up, , whichever occurred first.
Relapse free survival | up to 2 years after the date of the last enrolled participants
  The interval from CR to the date of relapse, or the date of death, or the date of last follow-up, whichever occurred first. This outcome analyzes patients achieved CR in two courses of induction therapy.
30-day mortality | Within 30 days of the date of the last enrolled participants
  Percentage of patients who died within 30 days from enrollment
60-day mortality | Within 60 days of the date of the last enrolled participants
  Percentage of patients who died within 60 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, doctor, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang ES, Goldberg AD, Tallman M, Walter RB, Karanes C, Sandhu K, Vigil CE, Collins R, Jain V, Stone RM. Crenolanib and Intensive Chemotherapy in Adults With Newly Diagnosed FLT3-Mutated AML. J Clin Oncol. 2024 May 20;42(15):1776-1787. doi: 10.1200/JCO.23.01061. Epub 2024 Feb 7. PMID 38324741
- [Background] Department of Error. Lancet. 2023 Oct 14;402(10410):1328. doi: 10.1016/S0140-6736(23)02235-3. No abstract available. PMID 37838437
- [Background] Knight TE, Edwards H, Meshinchi S, Taub JW, Ge Y. "FLipping" the Story: FLT3-Mutated Acute Myeloid Leukemia and the Evolving Role of FLT3 Inhibitors. Cancers (Basel). 2022 Jul 13;14(14):3398. doi: 10.3390/cancers14143398. PMID 35884458